CLINICAL TRIAL: NCT03562572
Title: Ischemia (FFR) Driven Complete Revascularization Versus Usual Care in Patients With Non-ST Elevation Myocardial Infarction and Multivessel Diseases: The South Limburg Myocardial Infarction Study Group The SLIM Study
Brief Title: FFR Driven Complete Revascularization Versus Usual Care in NSTEMI Patients and Multivessel Disease
Acronym: SLIM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Collaborators: Maastricht University Medical Center (Other); Radboud University Medical Center (Other); Jeroen Bosch Ziekenhuis (Other); VieCuri Medical Centre (Other); Gottsegen György Országos Kardiológiai Intézet (Unknown); Bács-Kiskun County Teaching Hospital (Other); Brno University Hospital (Other); Szeged University (Other)
Responsible Party: Principal Investigator, Saman Rasoul, Principal Investigator, Zuyderland Medisch Centrum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-T-142; 28708 (Other: NTR)
Record Dates: First submitted 2018-05-23; First posted 2018-06-19 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease; NSTEMI - Non-ST Segment Elevation MI; Fractional Flow Reserve, Myocardial; Myocardial Revascularization; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: It concerns an investigator initiated prospective 1:1 randomised clinical trial in non-STEMI patients with multivessel coronary artery disease amenable to treatment with PCI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ischemia driven revascularization (Experimental): In the ischemia driven complete revascularisation strategy group all flow limiting (FFR ≤ 0.80) lesions will receive treatment by PCI and stenting. The non-IRA PCI should be performed during the same intervention. Exceptions can be made for complex lesions where the operator estimates that the revascularisation procedure will require significant contrast overload, which may lead to deterioration of cardiac and renal function of the patient.
  Interventions: Procedure: Ischemia driven revascularization
- Usual care group (Active Comparator): In the randomised to usual care group the procedure will stop after the PCI of the culprit artery and the patient will be referred to his treating cardiologist and/ or heart team who will decide whether a staged PCI of the non- IRA artery should take place. If the treating cardiologist (after advise of the heart team) decides to perform the non-IRA PCI revascularisation, than such treatment should take place within six weeks from the primary PCI in order to count as a scheduled staged PCI procedure.
  Interventions: Other: Usual care group

INTERVENTIONS:
Procedure: Ischemia driven revascularization — In the ischemia driven complete revascularisation strategy group all flow limiting (FFR ≤ 0.80) lesions will receive treatment by PCI and stenting during the index intervention
  Arms: Ischemia driven revascularization
Other: Usual care group — In the randomised to usual care group the procedure will stop after the PCI of the culprit artery and the patient will be referred to his treating cardiologist and/ or heart team who will decide whether a staged PCI of the non- IRA artery should take place. If the treating cardiologist (after advise of the heart team) decides to perform the non-IRA PCI revascularisation, than such treatment should take place within six weeks from the primary PCI in order to count as a scheduled staged PCI procedure.
  Arms: Usual care group

SUMMARY:
To compare FFR guided complete revascularization during the index procedure with usual care in non-STEMI patients with multivessel disease.

DETAILED DESCRIPTION:
Background:

Patients with non-ST elevation myocardial infarction (non-STEMI), as compared with STEMI patients, have a higher risk profile, more often MVD and less favourable outcome. Recent studies showed that complete revascularization in STEMI patients is feasible and effective. However, there is no clear evidence regarding the role of complete coronary revascularization by PCI in patients with non-STEMI with MVD.

Objective:

To compare FFR guided complete revascularization during the index procedure with usual care in non-STEMI patients with multivessel disease.

Design:

Prospective, multicentre, 1:1 randomized, investigator initiated study.

Hypothesis:

FFR guided complete percutaneous revascularisation of all significant stenosis in the non-culprit lesion performed within the index PCI procedure will improve clinical outcomes compared to the usual care, guided by discretion of the physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18-85 years presenting with non-STEMI according to current guidelines, who will be treated with PCI of the culprit and have at least one stenosis of >50% in a non-IRA on QCA or visual estimation of baseline angiography and judged feasible for treatment with PCI by the operator.
* Non-IRA stenosis amenable for PCI treatment (operator's decision)
* Signed informed consent

Exclusion Criteria:

* Left main disease (stenosis > 50%)
* Chronic total occlusion of a non-IRA
* Indication for or previous coronary artery bypass grafting
* Uncertain culprit lesion
* Complicated IRA treatment, e.g. extravasation, permanent no re-flow after IRA treatment (TIMI flow 0-1) and inability to implant a stent
* Known severe cardiac valve dysfunction that will require surgery or TAVI in the follow-up period.
* Killip class III or IV during the completion of culprit lesion treatment.
* Life expectancy of < 1 year.
* Intolerance to Aspirin, Clopidogrel, Prasugrel, Ticagrelor or Heparin.
* Gastrointestinal or genitourinary bleeding within the prior 3 months.
* Planned elective surgical procedure necessitating interruption of thienopyridines during the first 6 months post enrolment.
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Estimated)
Dates: Start 2018-06-07 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
The incidence of MACE at 12 months | 12 months
  MACE = The composite endpoint of all cause death, non-fatal Myocardial Infarction, any revascularisation and stroke at 12 months.

SECONDARY OUTCOMES:
The incidence of MACE in subgroups at 12 and 24 months. | 12 and 24 months
  Prespecified subgroup analyses of primary outcomes will be performed for:
  1. Diabetic patients versus non-diabetic patients
  2. Elderly (≥ 75 years) versus young patients (< 75 years)
  3. Male versus Female gender
  4. High versus low risk patients according to GRACE Risk Score
  5. Patients previous myocardial infarction versus patients with no previous myocardial infarction
  The Global Registry of Acute Coronary Events (GRACE) score estimates the admission 6 month mortality for patients with acute coronary syndrome. The GRACE score ranges from 0 to > 285. A higher GRACE represents a higher mortality risk, ranging from 0-2% when the GRACE is between 0 and 87, to 99% when the GRACE exceeds 285.
Composite endpoint of Net Adverse Clinical Events (NACE) defined as composite endpoint of Cardiac death, Myocardial Infarction, any Revascularisation, Stroke and major bleeding at 12, 24 and 36 months. | 12, 24 and 36 months
Composite endpoint hospitalisation for heart failure and unstable angina pectoris at 12, 24 and 36 months. | 12, 24 and 36 months
All-cause mortality or Myocardial infarction at 12, 24 and 36 months. | 12, 24 and 36 months
Any revascularisation at 12, 24 and 36 months. | 12, 24 and 36 months
Stent thrombosis at 12, 24 and 36 months. | 12, 24 and 36 months
Bleeding (major and minor) at 48 hours and 12 months. | 48 hours and 12 months
The incidence of MACE at 36 months as well as outcomes of each component of MACE at 12 and 24 and 36 months. | 12, 24 and 36 months
  MACE = The composite endpoint of all cause death, non-fatal Myocardial Infarction, any revascularisation and stroke at 12 months.
Left ventricular ejection fraction at 12 and 24 and 36 month (MIBI scan, MRI or Echocardiography). | 12, 24 and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Saman Rasoul, Dr., Principal Investigator — Zuyderland MC; Arnoud van 't Hof, Prof. Dr., Study Director — Zuyderland MC
Locations (9):
- Brno University Hospital, Brno, Czechia
- Hungary (3):
  - Gottsegen György Országos Kardiológiai Intézet, Budapest
  - Bacs-Kiskun Teaching Hospital, Kecskemét
  - Szeged University, Szeged
- Netherlands (5):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Zuyderland MC, Heerlen
  - Maastricht University Medical Centre, Maastricht
  - Radboud University Medical Centre, Nijmegen
  - Viecuri Medisch Centrum, Venlo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pustjens TFS, Veenstra L, Camaro C, Ruiters AW, Lux A, Ruzsa Z, Piroth Z, Ilhan M, Vainer J, Gho B, Winkler PJC, Stein M, Theunissen RALJ, Kala P, Polad J, Berta B, Gabrio A, van Royen N, van 't Hof AWJ, Rasoul S. Fractional Flow Reserve-Guided Complete vs Culprit-Only Revascularization in Non-ST-Elevation Myocardial Infarction and Multivessel Disease: The SLIM Randomized Clinical Trial. JAMA. 2025 Nov 11;334(18):1628-1637. doi: 10.1001/jama.2025.16189. PMID 40886310